CLINICAL TRIAL: NCT04662658
Title: Hyperpolarized Xenon-129 MR Imaging of the Lung:E-cigarette Sub-study
Brief Title: Hyperpolarized Xenon-129 MR Imaging of the Lung
Acronym: e-cigarette
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Duke University (Other)
Responsible Party: Principal Investigator, Y. Michael Shim, MD, Medical Doctor, University of Virginia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 13740
Record Dates: First submitted 2020-11-02; First posted 2020-12-10 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: E-Cig Use
Keywords: e-cigarette use with young adults
MeSH Terms: conditions — Vaping | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups in parallel for the duration of the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Visit 1 UVA (Other): Visit 1 will last approximately 4 hours, and will include consenting, collection of data, questionnaires, and procedures as follows:
  1. Informed consent
  2. Demographic data
  3. Smoking history
  4. Medical history review
  5. Medication review
  6. Limited physical exam
  7. 6-minute walk test
  8. St. George's Respiratory Questionnaire (SGRQ)
  9. Baseline dyspnea index (BDI)
  10. Chronic respiratory questionnaire (CRQ)
  11. PFTs including:
      1. Pre-bronchodilator spirometry/ post bronchodilator spirometry.
      2. Body plethysmography (static lung volumes)
      3. Carbon monoxide diffusion capacity (DLCO)
  12. Collection of peripheral blood (20mL), exhaled breath condensate (EBC), and urine
  13. Hyperpolarized xenon-129 MRI (HXeMRI) if all eligibility criteria are met
  Interventions: Drug: Hyperpolarized Xenon -129 MRI
- Visit 2 Duke University (Other): Visit 2 will last about 3 hours, and will occur within 2-12 weeks of Visit 1. The purpose of this study visit is to obtain a measure of basic test-retest variability on 6 e-cigarette users and 6 control subjects. Participants will be selected based on age and sex matching needs at the time of enrollment.
  During Visit 2, changes in health since Visit 1 will be assessed. In addition, the following will be done in accordance with the parent protocol:
  1. The standard MR compatibility screening form will be completed.
  2. Spirometry will be performed before and after MR imaging.
  3. A limited physical exam
  4. Female subjects who could be pregnant will take a urine pregnancy test prior to imaging.
  5. Xenon MRI will be performed
  In addition to the above, the following will be completed:
  * Carbon monoxide diffusion capacity (DLCO)
  * Peripheral blood (20mL) and urine
  Interventions: Drug: Hyperpolarized Xenon -129 MRI

INTERVENTIONS:
Drug: Hyperpolarized Xenon -129 MRI — e-cigarette sub-study
  Other Names: MRI with xenon-129 gas

SUMMARY:
Over the past 10 years, electronic cigarettes (e-cigarettes, EC) have been commercialized as a "less harmful" alternative to traditional cigarettes.1,2 However, e-cigarettes are believed to cause pulmonary epithelial, endothelial and vascular dysfunction, and to cause murine phenotypes similar to those of human COPD. Recently, "spiked" vape juice has been linked to severe lung damage. Unfortunately, the effects of e-cigarettes on the human lungs are still poorly understood, especially in healthy young adults. Therefore, establishing the health effects of e-cigarettes in humans is of paramount importance to guide medical and regulatory decision making. Its widespread use and immense popularity among teenagers and young adults have caused major concern given potentially significant addictive and detrimental long-term health effects.

DETAILED DESCRIPTION:
This exploratory proposal will exploit 3D hyperpolarized xenon-129 MRI (HXeMRI), an imaging tool that our research group has pioneered, to address this urgent need. The HXeMRI technique has unique abilities to quantify regional ventilation (airflow), and gas uptake by tissue (interstitium), and blood (pulmonary vasculature) in the human lung with high spatial resolution. HXeMRI is anticipated to overcome the limitations of PFT and MDCT. Because HXeMRI images are acquired in a single breath-hold, pixel-based ratio maps can quantify xenon movement crossing from airways to tissue and finally to RBCs. The calculated ratios are closely related to important lung physiological factors: Tissue-to-Gas ratio (T/G) reflects tissue integrity and alveolar surface-to-volume ratio; RBC-to-Gas ratio (R/G) reflects overall gas exchange efficiency from the airspaces to the blood, and RBC-to-Tissue ratio (R/T) reflects capillary perfusion and gas-blood barrier functional integrity. The sensitivity and specificity of these parameters have been shown to be highly relevant in clinical arenas. For example, decreases in gas uptake by tissue and blood are consistently found in COPD and interstitial lung disease. Alteration of gas exchange measured by RBC-to-tissue ratio in COPD and asthma is associated with changes in the alveolar septal wall and capillary perfusion. Investigators have found regionally heterogeneous tissue gas uptake and impairment of gas exchange in idiopathic pulmonary fibrosis. This actively-funded NIH study has found highly heterogeneous airway obstruction and alterations of gas exchange in patients with cystic fibrosis that are routinely undetectable by clinical PFT. These results demonstrate the unique advantages of HXeMRI to quantitatively assess comprehensive regional physiology of microscopic pulmonary compartments.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects 21-30 years of age
2. At baseline health with no recent illnesses or medical conditions that would preclude enrollment as assessed by the Principal Investigator
3. Ability to understand a written informed consent form and comply with the requirements of the study.
4. E-cigarette use for more than 6 months preceding the date of enrollment and less than a 5 pack year smoking history (e-cigarette users) OR less than a 5 pack year smoking history (non-smoker group).
5. No diagnosis of any lung disease (pre-bronchodilator FEV1/FVC normal on the day of screening defined by > 95thCI of NHANES III, ATS/ERS guideline)

Exclusion Criteria:

1. History of any lung disease
2. Control (non-smoking) group: History of illegal drug use by inhalation
3. History of CNS disease including stroke and dementia, end-stage liver disease, coronary artery disease, renal failure
4. Acute infection of any kind in the previous 6 weeks
5. Pregnancy or a possibility of pregnancy
6. Anemia
7. Inability to undergo MR imaging based on the standard clinical criteria for MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-11-05 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Hyperpolarized xenon-129 MRI of the lung: e-cig sub-study | 12 months
  To measure the pulmonary physiologic effects of e-cigarette use in young adults with less than a 5 pack-year history of smoking traditional cigarettes.

CONTACTS AND LOCATIONS:
Overall Officials: Yun M shim, MD, Principal Investigator — University of Virginia
Locations (1):
- Snyder Building 480 Ray C. Hunt Drive, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No